CLINICAL TRIAL: NCT03915145
Title: Assistant Professor, Physioterapist, PhD
Brief Title: The Effects of Kinesio Taping in Women With Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, Assistant Professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 442-15
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio tape group (Experimental): Kinesio tape application has been applied
  Interventions: Other: Kinesio tape application
- Sham group (Sham Comparator): Sham kinesio tape application has been applied
  Interventions: Other: Sham Kinesio tape application
- Control group (Other): No intervention has been applied
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Kinesio tape application — Kinesio tape application will be performed.Taping is carried out from the estimated day of ovulation (cycle length in days minus 14) until the next menstrual period begins
  Arms: Kinesio tape group
Other: Sham Kinesio tape application — Sham kinesio tape application will be performed. Sham taping is carried out from the estimated day of ovulation (cycle length in days minus 14) until the next menstrual period begins
  Arms: Sham group
Other: No intervention — The natural process will be followed from the estimated day of ovulation (cycle length in days minus 14) until the next menstrual period begins
  Arms: Control group

SUMMARY:
The aim of our study was to investigate the effects of kinesio taping in women with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years of age,
* having Primary Dysmenorrhea
* being volunteer women

Exclusion Criteria:

* having give birth,
* having a serious psychiatric disorder
* having used oral contraceptive or depression drug in the last 6 month
* having secondary dysmenorrhea
* having irregular menstrual cycle
* having allergy to taping

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The severity of menstrual pain assessed with Visual Analog Scale | An average of 2 weeks
  A 10-cm Visual Analog Scale anchored from zero (no pain at all) to 10 (the worst pain I have ever felt) was used to determine the severity of each subject's menstrual pain.

SECONDARY OUTCOMES:
The complaints related to menstruation will be evaluated by a form prepared by the researchers | An average of 2 weeks
  The form assessing the complaints related to menstruation will be evaluated existing complaints affect the patient and expressed as, no, little, mederate, very.
The level of anxiety will be evaluated with The Spielberger State Trait Anxiety Inventory | An average of 2 weeks
  The Spielberger State Trait Anxiety Inventory is a 40-item self-report inventory designed to measure both state anxiety section (current feelings of apprehension, worry, etc.) and trait anxiety section (continuous feelings of apprehension, worry, etc.). Each section is scored on four levels of anxiety intensity from 1="not at all" to 4="very much" and with a sum score between 20 and 80. A higher total score indicates more severe anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda TOPRAK CELENAY, Principal Investigator — Ankara Yildirim Beyazıt University; Basak Kavalci, Study Chair — Gümüşhane Universıty; Aysenur Karakus, Study Chair — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)